CLINICAL TRIAL: NCT01065129
Title: A Phase I Trial Evaluating the Effects of Plerixafor (AMD3100) and G-CSF in Combination With Azacitidine (Vidaza) for the Treatment of MDS
Brief Title: Plerixafor and Granulocyte Colony-stimulating Factor (G-CSF) in Combination With Azacitidine for the Treatment of Myelodysplastic Syndrome (MDS)
Acronym: MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0150 / 201101810
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; plerixafor; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Level 1 (Experimental): AMD3100 320 μg/kg SC Days 1-5 of each 28 day cycle.
  Azacitidine 75 mg/m2 SC Days 1-5 of each 28 days cycle.
  G-CSF 5 μg/k SC Days 1-5 of each 28 days cycle.
  Interventions: Drug: G-CSF; Drug: Plerixafor; Drug: Azacitidine
- Dose Level 2 (Experimental): AMD3100 440 μg/kg SC Days 1-5 of each 28 day cycle.
  Azacitidine 75 mg/m2 SC Days 1-5 of each 28 days cycle.
  G-CSF 5 μg/k SC Days 1-5 of each 28 days cycle.
  Interventions: Drug: G-CSF; Drug: Plerixafor; Drug: Azacitidine
- Dose Level 3 (Experimental): AMD3100 560 μg/kg SC Days 1-5 of each 28 day cycle.
  Azacitidine 75 mg/m2 SC Days 1-5 of each 28 days cycle.
  G-CSF 5 μg/k SC Days 1-5 of each 28 days cycle.
  Interventions: Drug: G-CSF; Drug: Plerixafor; Drug: Azacitidine
- Expanded DLT Cohort (Experimental): After the MTD is determined, patients will be enrolled at the MTD dose of plerixafor. These patients will not receive G-CSF priming but will be treated with plerixafor and azacitidine for 2 cycles.
  Interventions: Drug: Plerixafor; Drug: Azacitidine

INTERVENTIONS:
Drug: G-CSF
  Other Names: Neupogen; Filgrastim
  Arms: Dose Level 1; Dose Level 2; Dose Level 3
Drug: Plerixafor
  Other Names: Mozobil
Drug: Azacitidine
  Other Names: Vidaza; 5-azacytidine

SUMMARY:
Our main objectives are to determine the optimal dose and schedule of plerixafor + G-CSF and azacitidine in patients with MDS and determine the safety and tolerability of plerixafor + G-CSF and azacitidine.

DETAILED DESCRIPTION:
The interaction of normal stem cells with the bone marrow microenvironment is mediated by a number of factors. These interactions have been implicated in protecting malignant hematopoietic cells from spontaneous apoptosis and genotoxic stresses such as chemotherapy. Key elements are CXCR4, which is expressed on normal stem cells and leukemic blasts, and its ligand, stromal derived factor 1 (SDF-1) expressed by bone marrow stromal cells and osteoblasts. The CXCR4/SDF-1 axis is essential for homing, retention and mobilization of stem cells from the bone marrow microenvironment. Plerixafor is a bicyclam small molecule inhibitor of CXCR4 and has been extensively studied by our group and others as a potent stem cell mobilization agent both in combination with G-CSF or alone (25, 62). Plerixafor is currently being investigated in a phase I/II trial in combination with salvage chemotherapy for relapsed AML in an attempt to sensitize leukemia stem cells to chemotherapy. The goal of this study is to determine the optimal dose of plerixafor for the treatment of patients with high-risk myelodysplastic syndrome (MDS) in combination with G-CSF and azacitidine. We hypothesize that plerixafor in combination with G-CSF will detach MDS blasts from the bone marrow microenvironment resulting in their increased proliferation and sensitivity to azacitidine; thus, improving complete and partial response rates (CR/PR).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed MDS with 5-20% blasts on bone marrow aspirate at the time of study enrollment AND at least one cytopenia.
* MDS is defined by the WHO criteria
* Previous therapy with decitabine or azacitidine will be allowed but patients must be at least 4 weeks from prior chemotherapy or radiation.
* Age >=18 years. Because no dosing or adverse event data are currently available on the use of plerixafor in combination with G-CSF or azacitidine in patients <18 years of age, children are excluded from this study; however, they will be eligible for future pediatric phase II combination trials.
* Life expectancy of greater than 2 months.
* ECOG performance status <= 2 (Karnofsky >=60%; see Appendix 1).
* Patients must have normal organ function as defined below:
* total bilirubin ≤ 1.5 X institutional upper limit of normal
* AST ≤ 2.0 X institutional upper limit of normal
* creatinine within normal institutional limits OR
* creatinine clearance >=60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Ability of the patient (or legally authorized representative, if applicable) to understand and the willingness to sign a written informed consent document.
* Females of child bearing potential must agree to abstain from sexual activity or to use a medically approved contraceptive measure/regimen during and for 3 months after the treatment period. Women of child bearing potential must have a negative serum or urine pregnancy test at the time of enrollment. Acceptable methods of birth control include oral contraceptive, intrauterine device (IUD), transdermal/implanted or injected contraceptives and abstinence. Males must agree to abstain from sexual activity or agree to utilize a medically approved contraception method during and for 3 months after the treatment period. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients with untreated 5q minus syndrome MDS
* Patients who have had G-CSF or GM-CSF within 2 weeks of the start of study
* Patients receiving any other investigational agents.
* Patients with known brain metastases. (These patients should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.)
* History of severe allergic or anaphylactic reactions attributed to compounds of similar chemical or biologic composition to plerixafor, azacitidine, G-CSF, or mannitol.
* History of sickle cell anemia. (G-CSF may initiate pain crises.)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because plerixafor, G-CSF, and azacitidine are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with azacitidine, G-CSF, or plerixafor, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with plerixafor. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients with advanced malignant hepatic tumors
* History of cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09-02 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2016-10-18 (Actual)

PRIMARY OUTCOMES:
Determine the optimal dose and schedule of plerixafor + G-CSF and azacitidine in patients with MDS | 42 days after the start of the second cycle of treatment
  The observation period for bone marrow aplasia as a DLT will be 42 days after the start of the second cycle of treatment or until the documentation of progression to leukemia.
  For all other toxicities, the DLT observation period will be 28 days from the start of treatment.
Determine the safety and tolerability of plerixafor + G-CSF and azacitidine | 30 days post-treatment

SECONDARY OUTCOMES:
Characterize the mobilization of MDS cells | Cycle 1 Day 5
Determine the pharmacokinetics of plerixafor on azacitidine | Cycle 1 Day 5
Determine progression free survival and response rates | 2 years
Freedom from transfusion | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schroeder, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu